CLINICAL TRIAL: NCT04004897
Title: Evaluation of Intracranial Pressure With Optic Nerve Sheath Diameter Measurement in Women With or Without Preeclampsia
Brief Title: Optic Nerve Sheath Diameter in Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Huseyin Kiyak, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Huseyin3
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preeclampsia group (Other): Patients with preeclampsia will receive optic nerve sheath diameter measurement with a linear ultrasound probe carefully and gently placed on the closed upper eyelids of patients.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement
- Pregnants without preeclampsia (Other): Pregnant women without preeclampsia will receive optic nerve sheath diameter measurement with a linear ultrasound probe carefully and gently placed on the closed upper eyelids of patients.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter measurement — Optic nerve sheath diameter measurement is performed with a linear ultrasound probe placed over the eyelid.

SUMMARY:
Severe preeclampsia is associated with an elevation in intracranial pressure (ICP). Optic nerve sheath diameter is a non-invasive surrogate of invasive ICP measurement. This study targets to evaluate the ICP in patients with or without preeclampsia.

DETAILED DESCRIPTION:
MRI studies have shown that brain edema due to an elevation in ICP develops in up to 70% of women with preeclampsia. Optic nerve sheath diameter is used to estimate the ICP and has been shown to correlate well with invasive ICP measurement. The present study aims to compare ICP using optic nerve sheath diameter in women with or without preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed as preeclampsia
* Age must be > 18 years

Exclusion Criteria:

* History of previous intracranial pathology or surgery
* Glaucoma

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
ICP | At 6th hour of admission
  The difference in ICP estimated with optic nerve sheath diameter measurement among women with or without preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Kiyak, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No